CLINICAL TRIAL: NCT03810222
Title: A Prospective Outcome Study in Patients With Moderate to Severe Traumatic Brain Injury in Bergamo Area (Italy)
Brief Title: A Prospective Outcome Study in Patients With Moderate to Severe Traumatic Brain Injury
Acronym: TBI-PRO
Status: Completed | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: TBI-PRO
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Brain Injuries, Traumatic; Brain Injury Traumatic Moderate; Brain Injury Traumatic Severe
Keywords: TBI moderate, TBI severe, GOSE
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: N/A (Observational Study) — This is an observational study and does not include interventions. Exposure is TBI.

SUMMARY:
Traumatic brain injury (TBI) is the leading cause of death, disability and cognitive impairment in young people worldwide. The majority of the traumatic deaths in developed countries results directly from lesions in the central nervous system. Furthermore, due to the persistence of disabling effects of TBI for many years, personal and public costs of supporting survivors have to be taken in consideration.

Many patients rescued by ICU treatment may have been severely disabled or vegetative because of trauma. These data suggest that, despite improvement in medical and surgical treatments, other factors related to trauma itself and to patient's condition could have an impact on the final outcome.

Aim of the TBI-PRO project is to collect high quality clinical and epidemiological data and to describe the outcome of moderate-to-severe TBI in a local contest (Bergamo area, Italy).

DETAILED DESCRIPTION:
All patients admitted to the ICU with a diagnosis of moderate-to-severe TBI, with or without polytrauma, are recruited. Bergamo hospital is the main Trauma Centre (Level I) and the only referring neurosurgical center within a population of 1.2 million inhabitants of Bergamo area. This hospital is also a Regional Pediatric Trauma Centre.

ELIGIBILITY:
Inclusion Criteria:

* admission to ICU
* diagnosis of moderate-to-severe TBI

Exclusion Criteria:

Patients who died in the first couple of hours after hospital admission are not included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the ICU with a diagnosis of moderate (Glasgow Coma Scale, GCS 9-13) or severe TBI (GCS 3-8), with or without associated polytrauma. Patients transferred from other hospitals within the first 24h are included.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale - Extended (GOSE) | 12 Months Post-Injury
  The global functional outcome at 12 months is assessed using the Glasgow Outcome Scale-Extended (GOS-E), obtained through structured interview. The GOS-E is a well-validated, widely employed measure of disability based on information on independence, employability, and social/community participation. The baseline function prior to injury is assessed to ensure that the deficit can be attributed to the event. GOS-E is dichotomized into favorable (a score of 5 to 8, Moderate Disability is defined by a score of 5-6) and unfavorable (a score of 1 to 4, Dead is defined by a score of 1).

SECONDARY OUTCOMES:
6-Month Outcome | 6 Months Post-Injury
  The functional outcome at 6 months is assessed using the GOS-E, neuroradiological findings (MRI Brain scan or CT) obtained within a 6 month-period post-injury are also considered.
Neuropsychological evaluation | 12 Months Post-Injury
  A neuropsychological test battery is designed to evaluate the cognitive domains commonly affected in survivors of moderate to severe TBI.

CONTACTS AND LOCATIONS:
Overall Officials: PAOLO GRITTI, MD, Principal Investigator — ASST- Papa Giovanni XXIII; FRANCESCO BIROLI, MD, Study Chair — Fondazione per la Ricerca Ospedale di Bergamo (FROM)
Locations (1):
- ASST- Papa Giovanni XXIII, Bergamo, Italy